CLINICAL TRIAL: NCT05982353
Title: Effect of Using a Hemostatic Gelatin Sponge Versus a Dense Polytetrafluorethylene Membrane for Socket Sealing Following Immediate Implant Placement. A Randomized Clinical Trial
Brief Title: Gelatin Sponge VS PTFE Membrane for Socket Sealing After Immediate Implant Placement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Alaa Emara, A.Professor OMFS, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTFEvsGelatin
Record Dates: First submitted 2023-07-30; First posted 2023-08-08 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Dental Implant Failed; Teeth Absent; Soft Tissue Injuries
Keywords: PTFE; immediate Implantation; Gelatin sponge; Dental socket
MeSH Terms: conditions — Anodontia; Soft Tissue Injuries | interventions — Gelatin Sponge, Absorbable

STUDY DESIGN:
Intervention Model Description: patients with dental sockets requiring immediate implantation with Gelatin Sponge vs polytetrafluoroethylene membrane
Who Masked: Participant
Masking Description: blinded envelopes selected by operator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PTFE application with immediate implantation (Sham Comparator): this group received PTFE membranes during immediate implantation as the gold standard
  Interventions: Device: PTFE application
- Gelatin Sponge application with immediate implantation (Experimental): this group received gelatin sponges during immediate implant placement
  Interventions: Device: Gelatin sponge

INTERVENTIONS:
Device: PTFE application — Polytetrafluoroethylene membrane used over immediate implants intraoperatively. Healing and osseointegration with the exposed membrane is assessed at the end of followup
  Arms: PTFE application with immediate implantation
Device: Gelatin sponge — gelatin sponge used over immediate implants intraoperatively. Healing and osseointegration with the exposed membrane is assessed at the end of followup
  Arms: Gelatin Sponge application with immediate implantation

SUMMARY:
Digital panoramas will be made to assess the implant sites. The included patients are assigned to their respective groups randomly. After implant submerging in the study group 2 layers of hemostatic resorbable gelatin sponge is fixed in the implant site; while with the control group PTFE is fixed. After 3 weeks the PTFE was removed while the gelatin sponge should be resorbed. 3 months later the implants are to be assessed for stability and a reverse torque test was used to confirm osseointegration during uncovering.

Follow-up appointments at 1,3 weeks and 1,2 & 3 months were planned.

DETAILED DESCRIPTION:
Dental implants are considered the gold standard for treatment of edentulous spaces. Immediate implant placement has multiple advantages including the shorter treatment span, less surgical procedures and faster loading possibility [1]. One of the drawbacks of immediate implant placement is proper soft tissue coverage of the submerged implant to prevent socket infection and allow implant stability and osseointegration [2]. To overcome these issues the use of membranes has been the standard procedure [3].

Polytetrafluoroethylene membranes (PTFE) have been reported vastly in literature and their results and clinical effect on soft tissue healing and guided tissue regeneration (GTR) around implants and in surgical sites. Dense PTFE allows for GTR by only promoting non-bacterial migration and improving cellular adhesion which promotes tissue regeneration underneath it [4]. On the other hand, PTFE membranes are quite expensive and with the economic crisis the world is facing the use of other less expensive options is crucial. Gelatin sponges are vastly used as hemostatic agents in minor surgical procedures and have shown excellent results in terms of hemostasis and rapid resorption [5]. The application of such material are multiple; such as with sinus lift procedures [6], microvascular decompression[7] and as a wound dressing [8].

The investigators hereby propose the use of hemostatic gelatin sponges as membranes for submerged immediate implants as a simpler and cheaper alternative to PTFE.

ELIGIBILITY:
Inclusion Criteria:

* patients with badly broken down tooth indicated for immediate implantation
* generally healthy patients 22-50 years of age
* non smokers
* good oral hygiene

Exclusion Criteria:

* poor bone quality
* poor oral hygiene
* non compliant patient

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
reverse torque test | 3 months after implant placement
  the implants will be subjected to a reverse torque test of 30 N/cm using a calibrated torque wrench. this should identify proper osseointegration.

SECONDARY OUTCOMES:
Clinical soft tissue healing | 2,3 weeks and 3 months
  incidence of infection/ improper tissue closure/dehiscence. will be assessed by to different blinded investigators using the Inflammatory Proliferative Remodeling scoring scale

CONTACTS AND LOCATIONS:
Overall Officials: Noha ElAdl, PhD, Study Director — National Research Centre, Egypt
Locations (1):
- National Research centre, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buser D, Chappuis V, Belser UC, Chen S. Implant placement post extraction in esthetic single tooth sites: when immediate, when early, when late? Periodontol 2000. 2017 Feb;73(1):84-102. doi: 10.1111/prd.12170. PMID 28000278
- [Background] Araujo MG, Silva CO, Souza AB, Sukekava F. Socket healing with and without immediate implant placement. Periodontol 2000. 2019 Feb;79(1):168-177. doi: 10.1111/prd.12252. PMID 30892762
- [Background] El Helow K, El Askary Ael S. Regenerative barriers in immediate implant placement: a literature review. Implant Dent. 2008 Sep;17(3):360-71. doi: 10.1097/ID.0b013e3181813406. PMID 18784536
- [Background] Carbonell JM, Martin IS, Santos A, Pujol A, Sanz-Moliner JD, Nart J. High-density polytetrafluoroethylene membranes in guided bone and tissue regeneration procedures: a literature review. Int J Oral Maxillofac Surg. 2014 Jan;43(1):75-84. doi: 10.1016/j.ijom.2013.05.017. Epub 2013 Jun 28. PMID 23810680
- [Background] Sharifi S, Maleki Dizaj S, Ahmadian E, Karimpour A, Maleki A, Memar MY, Ghavimi MA, Dalir Abdolahinia E, Goh KW. A Biodegradable Flexible Micro/Nano-Structured Porous Hemostatic Dental Sponge. Nanomaterials (Basel). 2022 Sep 30;12(19):3436. doi: 10.3390/nano12193436. PMID 36234564
- [Background] Sohn DS, Moon JW, Moon KN, Cho SC, Kang PS. New bone formation in the maxillary sinus using only absorbable gelatin sponge. J Oral Maxillofac Surg. 2010 Jun;68(6):1327-33. doi: 10.1016/j.joms.2010.02.014. PMID 20493382
- [Background] Chang B, Tang Y, Wei X, Li S. A New Application of Gelatin Sponge in the Treatment of Hemifacial Spasm by Microvascular Decompression: A Technical Note. J Neurol Surg A Cent Eur Neurosurg. 2022 Mar;83(2):183-186. doi: 10.1055/s-0040-1720994. Epub 2021 May 19. PMID 34010981
- [Background] Chanu NR, Bhattacharya K, Marbaniang D, Pal P, Ray S, Mazumder B. Evaluation of a novel melatonin-loaded gelatin sponge as a wound dressing. J Vasc Nurs. 2022 Mar;40(1):2-10. doi: 10.1016/j.jvn.2021.09.004. Epub 2021 Oct 20. PMID 35287830